CLINICAL TRIAL: NCT01619202
Title: Comparison of Driving Performance Among Trained and Untrained Novice Drivers: Validation of a Multidimensional Simulated Driving Assessment
Brief Title: Comparing Driving Performance Among Trained and Untrained Drivers Using a Driving Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Pennsylvania Department of Health (Other Government); National Institute of Nursing Research (NINR) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-009288; K99NR013548 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-14 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Prevention Harmful Effects; Accidents, Traffic; Accident Prevention
Keywords: accident prevention; Adolescent; examination, automobile driver; Driving simulator; Young drivers; Driving education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risk Anticipation-Perception Training (Experimental): Complete the Risk Anticipation-Perception Training (RAPT) program
  Interventions: Behavioral: Risk Anticipation -Perception Training
- No training program (No Intervention): Does not complete the Risk Anticipation-Perception Training (RAPT) program

INTERVENTIONS:
Behavioral: Risk Anticipation -Perception Training — Web-based computer training program designed to teach novice teen drivers how to properly scan for hazards
  Other Names: RAPT
  Arms: Risk Anticipation-Perception Training

SUMMARY:
The purpose of this study is to examine differences in driving performance on a simulated driving assessment between novice teen drivers who receive the Risk Anticipation-Perception Training (RAPT) program and novice teen drivers who do not receive the training program.

DETAILED DESCRIPTION:
Motor vehicle crashes remain the number one cause of death among teens in the United States. Teen drivers (ages 16 to 19) are four times more likely to be involved in fatal crashes than adult drivers (ages 25 to 69). Driving simulators are a safer alternative to on-road assessments that are often affordable and can provide experimental control for research. Though driving simulators have advantages for evaluating driving performance in teens, there are gaps in the literature on the validity of a multidimensional outcome of driving performance in a simulator. To further examine the validity of a multidimensional measure of driving performance in a simulator, we compare simulated driving performance among teens who are trained hazard anticipation-perception training and those who are not.

ELIGIBILITY:
Inclusion Criteria:

* Holds a valid driver's license for less than or equal to 180 days
* 16 - 18 years of age

Exclusion Criteria:

* Self-reports claustrophobia, migraine headaches, and/or motion sickness
* Females who are pregnant
* Previously participated in another CHOP driving simulator study
* Non-English Speaking

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Simulated driving performance measured by the number of errors made or the lack thereof, during a series of simulated drives. | at least 1 week after training or enrollment
  Simulated driving performance will be measured by the number of driving errors made during the simulated drives. The simulated driving performance will be compared across each arm, Intervention and Control. Intervention arm: Simulated driving performance will be measured at least 1 week after completion of the RAPT (Hazard Awareness) training program; Control arm: Simulated driving performance will be measured after enrollment and completion of pre-assessment measures.

CONTACTS AND LOCATIONS:
Overall Officials: Flaura K Winston, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States